CLINICAL TRIAL: NCT05288608
Title: Patient- Reported Outcomes After Fast Same-day Delivery of Palliative Radiotherapy Without Planning CT Using an Adaptive Delivery Platform (FAST-METS)
Brief Title: Evaluation of Fast, Same-day Delivery of Palliative Radiotherapy Without a Planning CT (FAST-METS)
Acronym: FAST-METS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Suresh Senan, Principal Investigator, Clinical professor, Amsterdam UMC, location VUmc
Other Study IDs: 2021.0568
Record Dates: First submitted 2022-02-28; First posted 2022-03-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simple palliation: Treatment of patients who are referred for palliative radiotherapy to uncomplicated metastases.
- Complex palliation: Treatment of patients who require treatment to a site of previous radiation, patients undergoing concurrent systemic therapy, and those requiring a radiation dose exceeding 8 Gy.

SUMMARY:
Palliative radiotherapy is an effective treatment for patients with painful bone metastases. Standard workflows often involve long waiting times or multiple visits. Fast palliation completed during a single clinic visit can be achieved by omitting a planning CT scan, and using available diagnostic imaging for treatment planning. The adaptive treatment platforms provides the possibility to adapt positions differences between the diagnostic CT and radiotherapy treatment of the target and organs at risk. In this study, the investigators will investigate the experiences of patients who have been treated with this fast-adaptive workflow (FAST-METS) using 2 questionnaires.

DETAILED DESCRIPTION:
Palliative radiotherapy is an effective treatment for patients with painful bone metastases, and currently the investigators have clinically implemented the FAST-METS procedure at the department. All patients referred for palliative radiotherapy, in whom diagnostic imaging performed within 4 weeks is available, are eligible for this adaptive workflow. Consultation by telephone is done beforehand to verify whether the complaints correspond to the location of the metastasis.

This single-institutional, explorative study will investigate the experiences and quality of life of patients who were treated with this workflow. Two study questionnaires are used, and informed consent will be obtained for both. The EQ-5D-5L questionnaire will be completed on the day of treatment, after 6 weeks and 3 months post-treatment. The other questionnaire used was developed for patients treated with adaptive radiotherapy. Two patients groups will be studied, namely those undergoing simple and complex palliative radiotherapy. Patients treated with complex palliative radiotherapy are defined as those referred for re-irradiation to the site of metastasis, patients undergoing concurrent systemic therapy, and patients treated with a single fraction radiation dose exceeding 8 Gy.

In addition, the study will evaluate time spent on treatment preparation and delivery proces, and dosimetric aspects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for palliative radiotherapy to metastases
* Recent diagnostic CT scan (preferably <4 weeks) of the metastasis with full body contour of the patient included.

Exclusion Criteria:

* A solitairy metastasis from a primairy tumor with good a prognosis
* A metastasis located in ventral ribs where respiratory motion of the target is expected
* Patients who are not fluent in Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for palliative radiotherapy, in whom diagnostic imaging performed in the preceding 4 weeks is available.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-12-16 (Estimated); Study Completion 2023-03-16 (Estimated)

PRIMARY OUTCOMES:
Quality of life of patients | 3 months
  Quality of life, with EQ-5D-5L questionnaires. The questionnaires comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Satisfaction of patients | 1 week
  Measure the satisfaction of patients who are treated with FAST-METS workflow, using a patient questionnaire developed in-house, which is completed on the day of treatment. Each question has 5 levels: not satisfied at all, some satisfaction, reasonably satisfied, and very satisfied

SECONDARY OUTCOMES:
Dosimetric data | 1 week
  Dosimetric data on treatment planning, containing volumes of gross tumor volume (GTV), planning target volume (PTV), coverage of GTV and PTV, dose to the organs at risk (OARs), technique of radiotherapy (IMRT/VMAT) and number of monitor units (MU). The data of the reference plan and the adapted plan will be collected and compared
Time spent on treatment preparation and delivery proces | 1 week
  The time spent in minutes at each step of the patient's treatment journey will be recorded, commencing from the start of clinical consultation until the patient leaves the radiotherapy department.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. Suresh Senan, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc, Department Radiation Oncology
Locations (1):
- AmsterdamUMC, location VUmc, Amsterdam, Netherlands